CLINICAL TRIAL: NCT00323050
Title: Evaluate Immunogenicity,Safety & Reactogenicity of a Booster Dose of Hib-MenC Conjugate Vaccine When Given to Healthy Subjects Aged 13-14 Months Who Were Primed With 3 Doses of Hib-MenC vs a Booster Dose of Infanrix Hexa Given to Subjects Primed With 3 Doses of Infanrix Hexa and Meningitec
Brief Title: Study of a Booster Dose of Hib-MenC Conjugate Vaccine vs Infanrix Hexa When Given to 14 Month Old Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 102547
Record Dates: First submitted 2005-08-26; First posted 2006-05-09 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Neisseria Meningitidis; Haemophilus Influenzae Type b
MeSH Terms: conditions — Haemophilus Infections | interventions — Vaccines

INTERVENTIONS:
Biological: Haemophilus influenzae type b- and meningococcal (vaccine)

SUMMARY:
The purpose of this study is to evaluate the immunogenicity, safety and reactogenicity of a booster dose of the Hib-MenC conjugate vaccine when given to healthy subjects aged 13 to 14 months who were primed with three doses of Hib-MenC compared to a booster dose of Infanrix hexa given to subjects primed with three doses of Infanrix hexa and Meningitec.

DETAILED DESCRIPTION:
The study is open and Infanrix hexa will serve as active control. Subjects will receive one vaccine dose of either Hib-MenC or Infanrix hexa, and will have 2 blood samples taken: before and one month after vaccination. Subjects who will receive a booster dose of Hib-MenC were primed with 3 doses of Infanrix penta + Hib-MenC or 2 doses of NeisVac-C and Infanrix hexa / Infanrix IPV/Hib.

ELIGIBILITY:
Inclusion criteria:

* Healthy male or female between, and including, 13 and 14 months of age
* Having participated in the primary vaccination study 217744/097.

Exclusion criteria:

* Previous vaccination against OR history of OR known exposure to diphtheria, tetanus, pertussis, hepatitis B, polio, H. influenzae type b (Hib) and/or meningococcal serogroup C disease except if within the framework of study 217744/097
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
* A family history of congenital or hereditary immunodeficiency
* History of any neurologic disorders or seizures

Ages: 13 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 468 (Actual)
Dates: Start 2004-11; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Percentage (%) of subjects with anti-PRP antibody concentrations (conc) ≥1µg/ml and % of subjects with SBA-MenC titers ≥ 128 one month post vaccination.

SECONDARY OUTCOMES:
Pre & 1M post vacc, S+/SP & conc/titer: SBA-MenC, anti-PSC,-PRP,-T & anti-PRP ≥ 1,-PSC ≥ 2, SBA-MenC ≥ 128
Pre vacc, S+/SP & conc/titer: anti-D,-PT,-FHA,-PRN,-HBs, -polio 1,2,3
Loc, gen sympt: D 0-3, unsol sympt: D 0-30 post vacc.
SAEs for whole study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- Spain (12):
  - GSK Investigational Site, Alcorcón
  - GSK Investigational Site, Almeira
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Basurto/Bilbao
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Getafe
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Móstoles/Madrid
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Valladolid
  - GSK Investigational Site, Vélez-Málaga

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 102547 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 102547 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 102547 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 102547 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 102547 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 102547 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register